CLINICAL TRIAL: NCT04849780
Title: Evaluation of Dryness in a Silicone Hydrogel Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6388
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ARM 1 (Experimental): Eligible subjects will be randomized to the TEST lens to wear in both eyes for approximately 2 weeks.
  Interventions: Device: ACUVUE Oasys 1-Day
- ARM 2 (Experimental): Eligible subjects will be randomized to the CONTROL lens to wear in both eyes for approximately 2 weeks. Then the subject will receive the TEST lens to wear in both eyes for approximately 2 weeks.
  Interventions: Device: ACUVUE Oasys 1-Day; Device: Habitual Lens

INTERVENTIONS:
Device: ACUVUE Oasys 1-Day — TEST
Device: Habitual Lens — Subjects' own Habitual Lenses
  Other Names: CONTROL
  Arms: ARM 2

SUMMARY:
This is a multi-site, randomized, bilateral, dispensing, parallel design study with two arms to evaluate contact lens related dry eye symptoms and subjective comfort.

ELIGIBILITY:
Inclusion Criteria:

- Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Between 18 and 59 (inclusive) years of age at the time of screening.
4. Be a daily disposable current soft contact lens wearer in both eyes with a minimum of 6 days/week wear time over the last 1 month by self-report.
5. Have a CLDEQ-8 score of 15 or greater with the habitual lens.
6. Subjects must possess a pair of spectacles for distance correction.
7. Subject's habitual lens must be the following lens types: Alcon DAILIES® Aqua Comfort Plus® , Alcon DAILIES TOTAL1®, CooperVision® clariti® 1 day, CooperVision® MyDay®, or Johnson & Johnson 1-Day ACUVUE® Moist.
8. The subject's vertex corrected spherical distance refraction must be in the range of -1.00 D to -6.00 D (inclusive) in each eye.
9. The magnitude of subject's vertex corrected refractive cylinder must be less than 1.00 diopter in each eye.

11. Have spherical best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

- Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Subject's habitual lens is ACUVUE OASYS®1-Day.
2. Currently pregnant or lactating, by self-report.
3. Any ocular or systemic allergies, disease or use of medication which may interfere with contact lens wear (at the discretion of the investigator).
4. Any active ocular abnormalities/conditions that may interfere with contact lens wear (at the discretion of the investigator).
5. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Habitual contact lens wear modality as extended wear (≥1 night per month of extended wear).
8. Habitual contact lens is rigid gas permeable, toric, monovision or multi-focal.
9. . Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
10. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrollment.
11. Employee or employee's immediate family member of clinical site (e.g., Investigator, Coordinator, Technician).
12. Current habitual use of Restasis, Xiidra, ocular steroids, or any medication (Rx or over the counter (OTC)) that may interfere with contact lens wear (at the discretion of the investigator).
13. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
14. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (9):
- United States (9):
  - Vue Optical Boutique, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Sacco Eye Group, Vestal, New York
  - Procare Vision Centers, Granville, Ohio
  - Dr. David Ferris & Associates, Warwick, Rhode Island
  - Optometry Group Pllc, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 95 subjects were enrolled in this study. Of those enrolled, 47 were randomized to Arm1 and dispensed at least one study lens, while 45 subjects were randomized to Arm 2 and were dispensed at least 1 study lenses. All dispensed subjects in Arm 1 completed the study while only 39 of those dispensed in Arm 2 completed the study. A total of 6 subjects were discontinued from Arm 2.
Groups:
- Arm 2: Subjects randomized to this Arm were dispensed their habitual lenses A for approximately 2 weeks, then returned for follow-up evaluation. Subjects were then dispensed senofilcon A for approximately 2 weeks, then returned for follow-up evaluation and were exited from the study.
- Arm 1: Subjects randomized to this Arm were dispensed the senofilcon A for approximately 2 weeks, then returned for follow-up evaluation and were exited from the study.
Period: Period 1
Arm/Group | Arm 2 | Arm 1
Started | 45 | 47
Completed | 41 | 47
Not Completed | 4 | 0
Not completed — Covid-19 Related | 1 | 0
Not completed — Subject no longer meet eligibility criteria | 3 | 0
Period: Period 2
Arm/Group | Arm 2 | Arm 1
Started | 41 | 0
Completed | 39 | 0
Not Completed | 2 | 0
Not completed — Subject no longer meet eligibility criteria | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (8.14) | 34.0 (8.42) | 34.3 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 16 | 11 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  White | 45 | 45 | 90
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Comfort Score
Description: Comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The change from baseline was calculated as 2-week follow-up minus baseline. The average change from baseline was reported for each arm. the change from baseline ranges from -120 to 120 where higher change from baseline comfort scores indicates a more favorable performance.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that completed all required study visits without a major protocol deviation impacting a primary or secondary endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Arm 1: Subjects that wore the senofilcon A lens for 2-weeks and then exited the study.
- Arm 2 (Subjects' Own Contact Lens): Subjects that wore their habitual lenses for 2-weeks and then wore senofilcon A for 2-weeks and then exited the study.
Arm/Group | Arm 1 | Arm 2 (Subjects' Own Contact Lens)
Number analyzed (Participants) | 46 | 39
Units on a scale | 28.99 (26.766) | -0.29 (10.245)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 (Subjects' Own Contact Lens); Test type: Non-Inferiority — It was calculated that 80 participants randomized in a 1:1 fashion between the two arms would have at least 80% power to detect a 5 points difference in mean change from baseline overall comfort. Sample size was determined using a 2-sided Satterthwaite t-test assuming unequal variances with an alpha level of 5%. A non-inferiority margin of -5 points was used; Bootstrapping methods; Population Mean Difference = 29.279, 95% CI 2-sided [24.602 to 33.732] — Population Mean difference was calculated as Arm 1 minus Arm 2

2. Secondary Outcome: Change From Baseline CLDEQ-8 Score
Description: The CLDEQ-8 is a validated outcome measure for soft contact lenses wearers. It has been highly correlated with habitual baseline status and change in overall opinion when subjects are refit with contact lenses. A CLDEQ-8 total score of ≥12 is proposed to identify contact lens wearers who could benefit from clinical management of their contact lens related symptoms. A three-point change in CLDEQ-8 total scores has also been shown to be clinically important. This study will include the symptomatic subjects who will have a CLDEQ total score of ≥15. CLDEQ-8 scores range from 0 to 30 where, higher CLDEQ-8 score indicates more dry eye symptoms with respect to contact lens wear. The change is calculated as 2-week minus Baseline. The change from baseline CLDEQ-8 score ranges from -30 to 30 where lower change from baseline CLDEQ-8 scores indicate better performance. The average change in CLDEQ-8 for each arm was reported.
Time Frame: Up to 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Arm 1 | Arm 2 (Subjects' Own Contact Lens)
Number analyzed (Participants) | 46 | 39
Unit on a scale | -10.83 (6.631) | -1.23 (3.638)
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 (Subjects' Own Contact Lens); Test type: Non-Inferiority — Sample size was determined based on the primary hypothesis only. A non-inferiority margin of 3 points was used; Heterogeneous Mixed model analysis; The Kenward and Roger method was used for the denominator degrees of freedom; LS Mean = -10.7, 95% CI 2-sided [-12.7 to -8.6], Standard Error of Mean 1.03 — Mean difference was calculated as Arm 1 minus Arm 2 (subjects' own contact lens)

3. Secondary Outcome: Comfort Score
Description: Comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The average comfort score was reported for each group within Arm 2 only.
Time Frame: 2-Week Follow-up
Population: Subjects randomized to Arm 2 and completed all required study visits without a major protocol deviation impacting a primary or secondary endpoint.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Groups:
- Arm 2 (Senofilcon A); Arm 2 (Subjects' Own Contact Lens): Subjects that wore dispensed own contact lenses for 2-weeks and then dispensed senofilcon A for 2-weeks and then exited the study.
Arm/Group | Arm 2 (Senofilcon A) | Arm 2 (Subjects' Own Contact Lens)
Number analyzed (Participants) | 39 | 39
Unit on a scale | 55.88 (25.721) | 29.69 (13.849)
Statistical Analysis 1: Comparison: Arm 2 (Senofilcon A) vs Arm 2 (Subjects' Own Contact Lens); Test type: Non-Inferiority — Sample size was determined based on the primary hypothesis only. A non-inferiority margin of -5 points was used; Heterogeneous Mixed model analysis; The Kenward and Roger method was used for the denominator degrees of freedom; LS Mean = 25.9, 95% CI 2-sided [19.0 to 32.9], Standard Error of Mean 3.30 — Mean difference was calculated as Arm 2 (senofilcon A), minus Arm 2 (subjects' own contact lens)

4. Secondary Outcome: CLDEQ-8 Score
Description: The CLDEQ-8 is a validated outcome measure for soft contact lenses wearers. It has been highly correlated with habitual baseline status and change in overall opinion when subjects are refit with contact lenses. A CLDEQ-8 total score of ≥12 is proposed to identify contact lens wearers who could benefit from clinical management of their contact lens related symptoms. A three-point change in CLDEQ-8 total scores has also been shown to be clinically important. This study will include the symptomatic subjects who will have a CLDEQ total score of ≥15. CLDEQ-8 scores range from 0 to 30 where, higher CLDEQ-8 score indicates more dry eye symptoms with respect to contact lens wear. The average CLDEQ-8 for each arm was reported.
Time Frame: 2-Week Follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Arm 2 (Senofilcon A) | Arm 2 (Subjects' Own Contact Lens)
Number analyzed (Participants) | 39 | 39
Unit on a scale | 12.46 (6.078) | 21.18 (3.698)
Statistical Analysis 1: Comparison: Arm 2 (Senofilcon A) vs Arm 2 (Subjects' Own Contact Lens); Test type: Non-Inferiority — A non-inferiority margin of 3 points was used; Heterogeneous mixed model analysis; LS Mean = -8.5, 95% CI 2-sided [-10.1 to -7.0], Standard Error of Mean 0.75 — Mean difference was calculated as Arm 2 (senofilcon A) minus Arm 2 (subjects' own contact lens)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. For subject in Arm 1 their study duration was approximately 2-weeks while subjects in Arm 2 study duration was approximately 1-month.
Groups:
- Senofilcon A: Subjects that wore the senofilcon A lens in either Arm of the study.
- Nelfilcon A: Subjects that wore the nelfilcon A lens during the first period in Arm 2
- Delfilcon A: Subjects that wore the delfilcon A lens during the first period in Arm 2
- Somofilcon A: Subjects that wore the somofilcon A lens during the first period in Arm 2
- Stenofilcon A: Subjects that wore the stenofilcon A lens during the first period in Arm 2
- Etafilcon A: Subjects that wore the etafilcon A lens during the first period in Arm 2
Arm/Group | Senofilcon A | Nelfilcon A | Delfilcon A | Somofilcon A | Stenofilcon A | Etafilcon A
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/11 | 0/10 | 0/5 | 0/2 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/11 | 0/10 | 0/5 | 0/2 | 0/17
Other Adverse Events (participants affected / at risk) | 0/88 | 0/11 | 0/10 | 0/5 | 1/2 | 0/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Senofilcon A (N=88) | Nelfilcon A (N=11) | Delfilcon A (N=10) | Somofilcon A (N=5) | Stenofilcon A (N=2) | Etafilcon A (N=17)
Covid - 19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04849780/Prot_SAP_000.pdf